CLINICAL TRIAL: NCT05566574
Title: RP-3500 (ATRi) + External Beam Radiotherapy (EBRT) for the Palliative Treatment of Metastatic Disease
Brief Title: A Study of RP-3500 in Combination With Standard Radiation Therapy in People With Solid Tumor Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Repare Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-222
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor; Metastatic Cancer
Keywords: Palliative treatment; RP-3500 (ATRi); External Beam Radiotherapy (EBRT); 22-222
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Single arm, phase I/II trial to assess safety and tolerability of RP-3500 and palliative RT.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RP-3500 in Combination With Standard Radiation Therapy (Experimental): Patients with metastatic cancers with identified mutations in ATM will be enrolled. All patients will receive a standard palliative RT (4Gy x 5 fractions) on Days 1-5 in combination with RP-3500 on Days 1-5. In the first phase of the study, a 3+3 study design will be used to identify a safe dose of RP-3500 (starting at 80 mg QD) in combination with palliative RT.
  Interventions: Drug: RP-3500; Radiation: External Beam Radiotherapy (EBRT)
- Pilot subcohort (Experimental): The primary objective is to assess 6 month local control rate of patients of new metastatic lesions with pathogenic ATM who haves received prior RP-3500 and palliative RT.
  Interventions: Drug: RP-3500; Radiation: External Beam Radiotherapy (EBRT)

INTERVENTIONS:
Drug: RP-3500 — RP-3500 on Days 1-5.
Radiation: External Beam Radiotherapy (EBRT) — Palliative radiation therapy (4Gy x 5 fractions) to a metastatic site on Days 1-5

SUMMARY:
The purpose of this study is to test the safety of the study drug, RP-3500 when given in combination with palliative external beam radiotherapy (EBRT) to people who have metastatic solid tumor cancer with a mutation of the ATM gene. The study researchers will do tests to find the highest dose of RP3500 that causes few or mild side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy with at least one metastatic lesion amenable to radiotherapy. Bone, visceral, and soft tissue are eligible.
* Mutation in ATM (deleterious or VUS; somatic or germline; monoallelic or biallelic)

  * Note: Homozygous Deletion in the ATM gene will also be allowed
* ECOG performance status 0-2 or KPS equivalent
* Age ≥18 years
* Expected survival greater than 6 months
* Participant or Legally Authorized Representative (LAR) able to provide written informed consent
* Patients of reproductive potential must agree to practice an effective contraceptive method
* Ability to swallow capsules and retain oral medications
* Acceptable organ function at Screening, as evidenced by the following laboratory data:

  1. Serum creatinine ≤1.5 × upper limit of normal (ULN) or calculated creatinine clearance ≥60 mL/min using the Cockcroft-Gault equation or by 24-hour urine collection
  2. Total bilirubin ≤1.5 × ULN or <3.0 × ULN if known Gilbert's disease
  3. Serum albumin ≥2.5 g/dL
  4. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN unless liver metastases are present and thought to be a reason for AST/ALT elevation, in which case they must be ≤5 × ULN
* Acceptable hematologic function at Screening:

  1. No red blood cell or platelet transfusions or growth factors within 7 days of the first dose of RP-3500
  2. Hemoglobin ≥9.5 g/dL
  3. ANC ≥1700 cells/mm^3
  4. Platelet count ≥130,000 cells/mm^3
* Resolution of all toxicities of prior therapy or surgical procedures to baseline or Grade 1 (except for neuropathy, hypothyroidism requiring medication and alopecia can be resolved to Grade ≤2)
* Negative pregnancy test (serum or urine) for women of childbearing potential (WOCBP) at Screening and prior to first study drug. Non-WOCBP is defined as 1) adequate time of amenorrhea for > 12 months plus adequate FSH level or 2) surgically or anatomically infertile
* Male patients with female partners of childbearing potential and WOCBP must follow a contraception method (oral contraceptives allowed) at least as conservative as Clinical Trial Facilitation Group (CTFG) recommendations during their participation in the study. WOCBP must follow the recommendations until 6 months following last dose of study drug and male patients must follow the recommendations for 6 months following last dose of study drug. Male patients must also refrain from donating sperm during their participation in the study and for 6 months following last dose of study drug

Exclusion Criteria:

* Previous radiotherapy to the intended treatment site
* Prior therapy with an ATR or DNA-dependent protein kinase (DNA-PK) inhibitor
* Serious medical co-morbidities precluding radiotherapy
* Pregnant or breast-feeding women
* No other concurrent systemic therapy during the entire duration of protocol treatment. Patients can have other systemic treatments up until the start of protocol treatment. Patients can also have other systemic treatments after the completion of protocol treatments
* Known hypersensitivity to any of the ingredients of RP-3500
* Uncontrolled hypertension (systolic blood pressure [BP] ≥160 mmHg; diastolic BP ≥100 mmHg) despite adequate treatment prior to first dose of RP-3500
* Patients with active, uncontrolled bacterial, fungal, or viral infection, including hepatitis B virus (HBV), hepatitis C virus (HCV), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness. In equivocal cases, patients whose viral load is negative, may be eligible. HIV seropositive patients who are healthy and low risk for AIDS related outcomes could be considered eligible. Eligibility criteria for HIV positive patients should be evaluated and discussed, and will be based on current and past CD4 and T-cell counts, history (if any) of AIDS-defining conditions (eg, opportunistic infections), and status of HIV treatment
* Moderate or severe hepatic impairment (ie, Child-Pugh class B or C)
* History or presence of an abnormal ECG that is clinically significant in the investigator's opinion, including complete left bundle branch block, second- or third-degree heart block, or recent history of myocardial infarction that in the opinion of the investigator will pose an increased risk of rhythm abnormalities
* History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias such as structural heart disease (eg, severe left ventricular systolic dysfunction, left ventricular hypertrophy), coronary heart disease (symptomatic or with ischemia demonstrated by diagnostic testing), clinically significant electrolyte abnormalities (eg, hypokalemia, hypomagnesemia, hypocalcemia), or family history of sudden unexplained death or long QT syndrome
* Current treatment with medications that are well-known to prolong the QT interval
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol and/or follow-up procedures outlined in the protocol
* Patients who are receiving strong CYP3A inhibitors or inducers, P-gp inhibitors and/or BCRP inhibitors
* Patients with germline homozygous ATM mutations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Phase I - Safety and Tolerability of RP-3500 in combination with radiation therapy | 2 years
  by assessing the grade and frequency of adverse events and serious adverse events. A dose limiting toxicity (DLT) will be graded according to NCI CTCAE v5.0.
Phase II - Assess 6 month local control rate of patients with pathogenic ATM who received RP-3500 and palliative RT | 2 years
  Imaging per discretion of treating physician, and may include PET, CT and MRI imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lee, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activites), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center at Suffolk-Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm